CLINICAL TRIAL: NCT01018602
Title: A Phase II, Randomized, Double-blind, 2-arm Controlled Study to Evaluate Efficacy of the DPPIV-inhibitor Vildagliptin for Prevention of Type 2 Diabetes in Women With a Recent History of Insulin-requiring Gestational Diabetes
Brief Title: PINGUIN (Postpartum Intervention in Women With Gestational Diabetes Using Insulin)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut fur Diabetesforschung, Munich, Germany (Other)
Responsible Party: Prof. Dr. med. Anette-G. Ziegler, Institut fur Diabetesforschung, Munich, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 808040006
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Insulin-dependent Gestational Diabetes
MeSH Terms: interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vildagliptin (Active Comparator)
  Interventions: Drug: vildagliptin
- inactive pill without active agent (Placebo Comparator): participants receive an inactive pill without active agent, but undergo the same examinations, visits and tests as the group treated with vildagliptin.
  Interventions: Drug: inactive pill

INTERVENTIONS:
Drug: vildagliptin — 100 mg per day over 24 months
  Arms: vildagliptin
Drug: inactive pill — 1 pill per day over 24 months
  Arms: inactive pill without active agent

SUMMARY:
The aim of the study is to prove the efficacy of the oral intake of vildagliptin in a daily dose of 100 mg in scope of the development of type 2 diabetes in women with insulin dependent gestational diabetes in their last pregnancy not longer than 9 months after birth.

In this randomized, placebo-controlled, double-blinded clinical phase II study, 140 participants aged 18 years or older and an insulin dependent gestational diabetes in their last pregnancy should be included and treated with vildagliptin or placebo over 24 months, followed by a 12 months observation period. Exclusion criteria are pregnancy and lactation as well as a clinical overt diabetes or islet autoimmunity.

The null hypothesis is that there is no significant difference of diabetes incidence (according to ADA criteria 1997) in both groups.

Primary endpoint is the clinical manifestation of diabetes, secondary endpoints include the improvement of beta cell function (evaluable by C-peptide measurement) and of insulin sensitivity by the treatment with vildagliptin.

ELIGIBILITY:
Inclusion Criteria:

* women with insulin-dependent gestational diabetes during the last pregnancy
* < 9 months after delivery
* age 18 years or older
* contraception during intervention period (at least 24 months)

Exclusion Criteria:

* pregnancy or lactation
* GADA or IA-2A positivity
* clinical overt diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
development of type 2 diabetes mellitus by criteria of ADA 1997 | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institut fuer Diabetesforschung, Munich, Germany

REFERENCES:
- [Derived] Hummel S, Beyerlein A, Pfirrmann M, Hofelich A, Much D, Hivner S, Bunk M, Herbst M, Peplow C, Walter M, Kohn D, Hummel N, Kratzsch J, Hummel M, Fuchtenbusch M, Hasford J, Ziegler AG; PINGUIN Study Group. Efficacy of vildagliptin for prevention of postpartum diabetes in women with a recent history of insulin-requiring gestational diabetes: A phase II, randomized, double-blind, placebo-controlled study. Mol Metab. 2018 Mar;9:168-175. doi: 10.1016/j.molmet.2017.12.015. Epub 2018 Jan 3. PMID 29396374